CLINICAL TRIAL: NCT06941038
Title: Effect of Intravesical Chemotherapy on Disease Recurrence in Patients Undergoing Nephroureterectomy for Upper Urinary Tract Urothelial Carcinoma
Brief Title: Intraoperative vs. Postoperative Intravesical Epirubicin Instillation for Prevention of Bladder Recurrence in High-Risk Upper Urinary Tract Urothelial Carcinoma
Acronym: IEPBR
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Cagri Akpinar, M.D, Ankara Etlik City Hospital
Other Study IDs: E2-21-421
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer Recurrence; Intravesical Instillation; Upper Urinary Tract Carcinoma
Keywords: bladder cancer; bladder cancer recurrence; intravesical instillation; upper urinary tract carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Upper urinary tract urothelial carcinoma (UTUC) accounts for 5%-10% of urothelial malignancies, with up to 50% of patients developing bladder recurrence post-RNU. High-risk UTUC (≥pT2, high-grade, or N+ disease) necessitates aggressive management. Intravesical chemotherapy mitigates recurrence risk, yet optimal timing-intraoperative vs. postoperative-remains unclear. This study evaluates intraoperative epirubicin instillation during RNU compared to postoperative administration and no instillation.

ELIGIBILITY:
Inclusion Criteria:

* primary high-risk UTUC.

Exclusion Criteria:

* prior bladder cancer,
* low-risk UTUC (managed conservatively),
* metastatic disease,
* incomplete follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between intravesical chemotherapy administered intraoperatively or postoperatively and bladder recurrence. | 365 days from the first instillation

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Ankara 06800, Ankara, Turkey (Türkiye)